CLINICAL TRIAL: NCT01823705
Title: Gastric Electrical Stimulation (GES) for the Treatment of Obesity
Acronym: GES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Corporate Technologies and New Ventures (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Exilis-1
Record Dates: First submitted 2013-03-26; First posted 2013-04-04 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gastric Electrical Stimulation (GES) (Experimental): Gastric Electrical Stimulation (GES) therapy for the treatment of obesity.
  Interventions: Device: Exilis Implantable Gastric Electrical Stimulation (GES)

INTERVENTIONS:
Device: Exilis Implantable Gastric Electrical Stimulation (GES)
  Other Names: Exilis Implantable Gastric Electrical Stimulation

SUMMARY:
The purpose of this feasibility study is to provide safety data on the implantable Exilis gastric electrical stimulation (GES) system, to individually adjust stimulation parameters to levels that are comfortable for implanted subjects during chronic daily treatment, and to collect data on acute gastrointestinal function and food intake responses to GES during in-clinic testing.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 21-64 with BMI of 40-45 kg/m^2 or BMI 35-39.9 kg/m^2 with at least one obesity-related comorbidity, who have failed prior non-surgical weight loss attempts, and have been within 5% of their current weight for at least one year.
* If diabetic, subject has non-insulin-dependent type 2 diabetes mellitus diagnosed within the last 7 years, and has an HbA1c level less than 8%.
* If female and of child-bearing age, subject is not pregnant or lactating and is willing to use effective contraception for the duration of the study.
* Subject is willing and able to complete scheduled study visits, complete on-line lifestyle educational modules, and complete required procedures.

Exclusion Criteria:

* Subject has a history of medical, surgical, or psychiatric conditions that, in the opinion of the Investigators, would limit study participation or contraindicate implantation of the Exilis GES system. Examples includes cardiac abnormalities contraindicating surgical anesthesia, prior gastrointestinal surgery, gastrointestinal motility disorders, inflammatory bowel disease, a history of eating disorders, anticipated future need for magnetic resonance imaging, or allergies to food ingredients in study test meals.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-03-29 (Actual); Primary Completion 2017-01-13 (Actual); Study Completion 2017-01-13 (Actual)

PRIMARY OUTCOMES:
First-in-human experience with the Exilis System, including initial clinical feasibility and safety data, as well as data on device performance (e.g., recharge durations and intervals) and use conditions (e.g., stimulation amplitudes, lead impedances). | Duration of study
  Once adjudicated by the Adverse Events Advisory Committee (AEAC), all adverse events recorded during the study were tabulated and summarized by seriousness, intensity, and related. Device performance and use conditions where characterized by collecting data on amplitude settings and lead impedance recorded during device interrogations and conducted at each clinic visits. The data will be tabulated and summarized using descriptive statistics, but no hypotheses tests were pre-specified
To gain an understanding of what sensations, if any, subjects feel during GES treatment, and what level and type of sensations subjects find acceptable and comfortable during chronic daily treatment. | 4 weeks
  In-clinic sensory testing and telephone follow-up were collected during Amplitude Titration phase and will be summarized. No formal hypothesis testing were pre-specified. Fourt separate visits were conducted approximately weekly during the titration phase. The testing procedure was expected to be repeated twice during each visits; once in a fasted state and once in a fed state. Subjects were asked to rate exposure sensitive from 0 (none) to 5 (intense)

SECONDARY OUTCOMES:
Change in gastric emptying time across a pair of in-clinic measurements made with and without GES. | Screening, Week 26 and Week 52
  During the two GI function visits subjects completed the same set of acute tests on two separate days, once with GES On and once with GES Off. Treatment ordering was randomly assigned in a balanced fashion. Each testing visit was preceded by a one week GES Off washout period. The gastric emptying half time outcomes in the acute cross-over experiment will be analyzed using the repeated measures regression with fixed subject and test-day effects, with the model-based t-test for the difference in the marginal means of T1/2 across treatments being used for statistical inference.
Change in whether GES delivered with the Exilis System suppresses post-meal gastric contractile activity | 8 and 10 weeks
  Antral motility index outcomes in the acute cross-over experiment were analyzed using the repeated measures regression with fixed subject and test-day effects. The model-based t-test for the difference in the marginal means of the MI values across treatments will be used for statistical inference.
Change in post-meal plasma glucose and insulin concentrations | Baseline and 6 months
  Blood samples were collected in conjunction with the gastric emptying test meals to explore whether GES alters plasma levels of gut peptides involved in regulating food intake and body weight, including GLP-1, PP, and CCK.
Changes in coloric intake during a standardized ad libitum solid meal consumed in a controlled setting | 8 and 10 weeks
  During the GI function tests in the acute-cross over experiments subjects were fed a macaroni and cheese meal in a controlled setting. the meal was given at each GI function visit once with GES On and once with GES Off. The caloric intake was measured during the visit to determine whether the GES On would reduce meal intake.
Change in physiological parameters, medication usage, and psychometric assessment scores that occur during chronic daily GES treatment with the Exilis System. | Study duration
  The values of physiological measures, psychometric assessment questionnaire scores and changes in these values from the Screening visit baseline will be summarized by visit using descriptive statistics. Medications will be categorized by their primary indications for use, and the proportion of subjects taking medications in each category and the mean number of medications in each category per subject will be calculated at each visit and plotted over time. No formal hypothesis testing will be conducted.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Scottsdale, Arizona
  - Louisville, Kentucky
  - Nashville, Tennessee
- Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No